CLINICAL TRIAL: NCT02784236
Title: INTEGRATED IMPACT ASSESSMENT a Telemedicine Program in the Care of Patients With Diabetes Mellitus Type 1 Intensive Treatment With Multiple Daily Injections.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY TC MENARINI
Record Dates: First submitted 2016-05-24; First posted 2016-05-27 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Metabolic Impact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pre-post evaluation (Other): All patients undergo the condition of telemedicine.
  Interventions: Device: telemedicine

INTERVENTIONS:
Device: telemedicine — The study population corresponds to patients> 18 and <65 years with DM1 of> 1 year of evolution, and treated with MDI HbA1c> 7%. It is changing one group of subjects between two observation times due to any intervention in this case the addition of a tele

SUMMARY:
Prospective study of 6 months of evolution in people with type 1 diabetes with insulin multidose (MDI) and HbA1c> 7%. Patients were evaluated clinical, metabolic and psychological baseline and at 6 months, with a telematic visit at 3 months. We analyzed: glycemic control (HbA1c), glycemic variability (SD and MAGE), depressive symptoms (BDI-II), anxiety (STAI), treatment-related (DDS) distress, fear of hypoglycemia (FH-15), adhesion treatment (SCI-R), quality of life (DQOL) and treatment satisfaction (DTSQ) and the platform.

ELIGIBILITY:
Inclusion Criteria:

* Patients with DM1 plus 1 year of evolution.
* Age ≥18 and <65 years.
* HbA1c prior to study inclusion> 7%.
* MDI intensive insulin therapy in basal-bolus regimen.
* Patients candidates for telemonitoring. Approximately 50% of the patients should work with phone or tablet with Android operating system with active data rate to use wireless solution (bluetooth) OnLine MenaDiab® telemedicine. The remaining patients will work with the USB cable solution telemedicine MenaDiab® OnLine.
* Patients who have given written informed consent.

Exclusion Criteria:

* Treatment with ISCI.
* Chronic kidney disease, liver disease, thyroid dysfunction (hypothyroidism except properly treated and controlled).
* Pregnant or planning pregnancy.
* Diabetes mellitus type 2.
* Severe psychological disorders.
* Lack of cooperation (informed consent).
* Patients who are participating in other clinical studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To analyze the metabolic impact measured through HbA1c of a telemedicine program by MenaDiab® online platform in the care of patients with DM1. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: MARIA SOLEDAD RUIZ DE ADANA, MD phD, Principal Investigator — Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud
Locations (1):
- FIMABIS, Málaga, Malaga, Spain

IPD SHARING:
Plan to Share IPD: No